CLINICAL TRIAL: NCT05492643
Title: A Single Center, Open Label Clinical Study to Evaluate the Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine (SYS6006) as Heterologous Booster in Participants Aged 18 Years and Older Vaccinated With Inactivated SARS-CoV-2 Vaccine
Brief Title: The Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine (SYS6006) as Heterologous Booster in Participants Aged 18 Years and Older Vaccinated With Inactivated SARS-CoV-2 Vaccine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYS6006-007
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-07

CONDITIONS: SARS-CoV-2; Safety; Immunotoxicity
Keywords: SARS-CoV-2; Vaccine; Safety; Immunotoxicity
MeSH Terms: interventions — SYS6006 COVID-19 vaccine; Immunity, Cellular; Immunity, Humoral; Safety

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A：2 doses of inactivated SARS-CoV-2 vaccine (Experimental): Group A: will enrol 500 participants who have received 2 doses of inactivated SARS-CoV-2 vaccine according to national immunization planning, whose last dose was given at least 6 months ago. They will be given one dose of the study vaccine (SYS6006) after enrolment.
  Interventions: Biological: one dose of the study SARS-CoV-2 mRNA Vaccine (SYS6006); Other: Cellular Immunity; Other: Humoral Immunity; Other: Safety
- Group B：3 doses of inactivated SARS-CoV-2 vaccine (Experimental): Group B: will enrol 500 participants who have received 3 doses of inactivated SARS-CoV-2 vaccine according to national immunization planning, whose last dose was given at least 6 months ago. They will be given one dose of the study vaccine (SYS6006) after enrolment.
  Interventions: Biological: one dose of the study SARS-CoV-2 mRNA Vaccine (SYS6006); Other: Cellular Immunity; Other: Humoral Immunity; Other: Safety

INTERVENTIONS:
Biological: one dose of the study SARS-CoV-2 mRNA Vaccine (SYS6006) — all the 1000 participants enrolled will be given one dose of the study SARS-CoV-2 mRNA Vaccine (SYS6006)
Other: Cellular Immunity — the first 30 participants enrolled in each group will take extra blood samples for specific cellular immune response as measured by ELISpot.
Other: Humoral Immunity — the first 100 participants enrolled in each group will take extra blood samples for humoral immunity testing and laboratory examination.
Other: Safety — all the 500 participants enrolled will undergo safety observation

SUMMARY:
This study plans to enrol 1000 participants 18 years and above, with ≥10% participants ≥60 years old. According to SARS-CoV-2 vaccine vaccination history, they will be evenly divided into 2 groups, Group A and Group B.

Group A: will enrol 500 participants who have received 2 doses of inactivated SARS-CoV-2 vaccine according to national immunization planning, whose last dose was given at least 6 months ago. They will be given one dose of the study vaccine (SYS6006) after enrolment.

Group B: will enrol 500 participants who have received 3 doses of inactivated SARS-CoV-2 vaccine according to national immunization planning, whose last dose was given at least 6 months ago. They will be given one dose of the study vaccine (SYS6006) after enrolment.

The study is devided into two stages, the first stage will enrol 200 participants with 100 in Group A and 100 in Group B. They will undergo laboratory examination, immunogenicity observation and safety observation. The first 30 participants in each group will take extra cellular immune testing; the second stage will enrol the remaining 800 participants for safety observation.

DETAILED DESCRIPTION:
All participants: all the 1000 participants enrolled will undergo safety observation.

Immunogenicity Subgroup: the first 100 participants enrolled in group A will be assigned to Group A1; the first 100 participants enrolled in group B will be assigned to Group B1. Blood samples will be taken from Group A1 and Group B1 participants (200 in total) for humoral immunity testing and laboratory examination.

Laboratory examination include blood routine examination, urine routine test, blood biochemistry, coagulation, thyroid function, cardiac enzymes and troponin.

Humoral immunity testing include serum SARS-CoV-2 neutralizing antibody detection as measured by live virus and pseudovirus assay, S1 protein specific IgG binding antibody detection as measured by ELISA.

Cellular immunity Subgroup: the first 30 participants enrolled in Group A1 and Group B1 will take extra blood samples for specific cellular immune response (60 in total) as measured by ELISpot.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older;
2. Vaccinated with 2 or 3 doses of marketed inactivated SARS-CoV-2 vaccine according to national immunization planning, whose last dose was given at least 6 months ago;
3. Willing and able to comply with study requirements, and other study procedures within 6 months after vaccination;
4. Female participants or partners of male participants of childbearing potential: from the first day of last menstruation cycle to the day of enrolment, must had no sexual behavior with a male or had effective contraceptive methods without failure; voluntarily agree to maintain abstinent or use effective contraception with their partners until 6 months after vaccination;
5. Based on medical history enquiry, physical examination, and blood routine examination, the investigator judges the participants as in a healthy status; Participants with mild underlying disease (for example chonic diseases like diabetes/hypertension/hyperlipemia, etc.) must be in a stable state without exacerbation (no admission to hospital or no major adjustment to treatment regimen, etc.) for at least 3 months prior to enrollment in this study.
6. Understand the contents of the ICF and voluntarily sign it.

Exclusion Criteria:

* 1.Received any licensed SARS-CoV-2 vaccines other than inactivated SARS-CoV-2 vaccine).

  2.History of Severe Acute Respiratory Syndrome (SARS), or SARS-CoV-2 infections.

  3.History of allergy to any component of the study vaccine or history of severe allergic reaction to the vaccine or drug (including but not limited to anaphylaxis, allergic laryngeal oedema, anaphylactic purpura, thrombocytopenic purpura, or localized allergic necrosis (Arthus reaction)).

  4.Positive SARS-CoV-2 RT-PCR results. 5.Axillary temperature ≥37.3°C at enrolment or 24 hours prior to vaccination. 6.Had a history of Human Immuno-deficiency Virus(HIV) infection or positive HIV test result before enrolment.

  7.A history or family history of convulsions, epilepsy, encephalopathy and psychosis.

  8.Malignant tumors in the active phase, malignant tumors not receiving adequate treatment, malignant tumors at potential risk of recurrence during the study period.

  9.With severe or un-controllable cardiovascular disease, thrombotic disease, neurological disease, blood and lymphatic system disease, liver and kidney disease, respiratory system disease, metabolic, skeletal muscular disease and autoimmune disease.

  10.Congenital or functional splenic deficiency, complete or partial splenectomy for any reason.

  11.Prolonged (defined as more than 14 days) use of immunosuppressive or other immunomodulatory drugs (e.g., corticosteroids, ≥20 mg/d prednisone or equivalent; however, inhaled and topical steroids are permitted) within 6 months prior to the vaccine.

  12.Any other inactivated vaccines given within 7 days prior to the study vaccination, or live-attenuated vaccines within 14 days prior to the study vaccination.

  13.Have received immunoglobulin or other blood products within 3 months prior to enrollment or plan to receive them during the study period.

  14.Blood donation or blood loss ≥ 450 mL within 1 month prior to enrolment, or planned donation during the study period.

  15.Is currently in or intent to participate in another clinical study at any time during the conduct of this study.

  16.For Women of Childbearing Potential (WOCBP): with a positive urine pregnancy test before vaccination; pregnant or lactating; or have a plan to become pregnant within 6 months after enrolment. For male participants whose partner is WOCBP: whose partner has a plan to become pregnant within 6 months after her partner's enrolment.

  17.With a history of intramuscular injection contraindication. For example: diagnosed thrombocytopenia, and coagulation disorder or received anticoagulation therapy.

  18.Participants deemed unsuitable for participation in this study based on the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-13 (Actual); Primary Completion 2023-02-27 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 6 months
  * Solicited (local and systemic) adverse events (within 14 days after vaccination) and unsolicited adverse events (within 30 days after vaccination);
  * Serious Adverse Events (SAE) (within 6 months after vaccination);
  * Adverse events of special interest (AESI) (within 6 months after vaccination);
  * Abnormal laboratory examination (4 days after vaccination).
Primary Immunogenicity Endpoint | 6 months
  Geometric Mean Titer (GMT), Geometric Mean Increase (GMI), Seroconversion (SCR) of SARS-CoV-2 live virus neutralizing antibody (14 days, 30 days post vaccination)

SECONDARY OUTCOMES:
GMT、GMI、SCR of SARS-CoV-2 pseudovirus neutralizing antibody | 14 days, 30 days post vaccination
  1.To evaluate the immunogenicity of one dose of SYS6006 mRNA vaccine as heterologous booster in participants aged 18 years and older who have received 2 or 3 doses of inactivated SARS-CoV-2 vaccine as measured by pseudovirus neutralizing antibody.
GMT、GMI、SCR of SARS-CoV-2 S1 protein specific binding IgG antibody | 14 days, 30 days post vaccination
  2.To evaluate the immunogenicity of one dose of SYS6006 mRNA vaccine as heterologous booster in participants aged 18 years and older who have received 2 or 3 doses of inactivated SARS-CoV-2 vaccine as measured by S1 protein specific IgG binding antibody.
GMT、GMI、SCR of SARS-CoV-2 live virus, pseudovirus neutralizing antibody and S1 protein specific IgG antibody | 3 months, 6 months post vaccination
  3.To evaluate the immuno-persistency of one dose of SYS6006 mRNA vaccine as heterologous booster in participants aged 18 years and older who have received 2 or 3 doses of inactivated SARS-CoV-2 vaccine as measured by SARS-CoV-2 live virus neutralizing antibody, pseudovirus antibody and S1 protein specific IgG binding antibody.

OTHER OUTCOMES:
Ratio of positive cells excreting specific cytokines (IFN-γ, IL-2, IL-4) by Enzyme Linked Immunospot Assay (ELISpot) (14 days, 30 days, 3 months, 6 months post vaccination) | 6 months
  To evaluate the cellular immunity level of one dose of SYS6006 mRNA vaccine as heterologous booster in participants aged 18 years and older who have received 2 or 3 doses of inactivated SARS-CoV-2 vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghuan Wang, Principal Investigator — Wuhan University; Jianying Huang, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China